CLINICAL TRIAL: NCT05887674
Title: Shanghai Non-pharmacological Intervention for Mild Cognitive Impairment and Mild Alzheimer's Disease: Combined Low Inflammatory-index Diet, Physical Exercises, and Cognitive Training in Nursing Home
Brief Title: Shanghai Non-pharmacological Intervention for Mild Cognitive Impairment and Mild Alzheimer's Disease
Acronym: SIM-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Sinopharm Nursing Care Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RJNeuroBank-SIM2
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
Keywords: mild cognitive impairment; Alzheimer's disease; Diet; Physical exercise; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-domain intervention group (Experimental): Patients in this arm will receive multi-domain life-style intervention including low inflammatory-index diet, exercise, and cognitive training.
  Interventions: Behavioral: Diet intervention; Behavioral: Exercise; Behavioral: Cognitive training
- Exercise and cognitive training (Experimental): Patients in this arm will receive the intervention of exercise and cognitive training.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive training
- Standard health counseling at baseline (No Intervention): Patients in this arm will have their habitual diet and life style. No particular intervention or consultation would be provided.

INTERVENTIONS:
Behavioral: Diet intervention — Low inflammatory-index diet
  Arms: Multi-domain intervention group
Behavioral: Exercise — Guided muscle strength training and stretching exercises
  Arms: Exercise and cognitive training; Multi-domain intervention group
Behavioral: Cognitive training — Cognitive training will be implemented in person
  Arms: Exercise and cognitive training; Multi-domain intervention group

SUMMARY:
This study is a multicentre, randomized, double-blind, controlled trial that aims to investigate the efficacy of multi-domain life-style intervention including low inflammatory-index diet, exercise, and cognitive training in patients with mild cognitive impairment and mild Alzheimer's disease.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, controlled trial that aims to investigate the efficacy of multi-domain life-style intervention including low inflammatory-index diet, exercise, and cognitive training in patients with mild cognitive impairment and mild Alzheimer's disease. Patients who eligible to the inclusion criteria and ineligible to the exclusion criteria will be randomly assigned into three groups by a 1:1:1 ratio. Patients in first arm will receive multi-domain life-style intervention including low inflammatory-index diet, exercise, and cognitive training. Patients in the second arm will receive intervention of exercise and cognitive training. Patients in the third arm will receive regular health advice. We hypothesize that the multi-domain intervention will reduce impairment in the study group compared to the control group during the 2-year intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60-90 years
2. In accordance with the diagnostic criteria for "mild cognitive impairment due to Alzheimer's disease" or "mild Alzheimer's disease" from the National Institutes of Health National Institute on Aging-Alzheimer's Association (NIA-AA) (2011)
3. The Hamilton depression rating scale/17 edition (HAMD) total score≤10
4. Neurological examination: no obvious signs
5. Education: primary school (grade 6) or above and capacity to complete tests for cognitive ability
6. Capacity to give consent

Exclusion Criteria:

1. Other causes of cognitive decline: cerebrovascular disease, central nervous system infection, Creutzfeldt-Jakob disease, Huntington's and Parkinson's disease, Creutzfeldt-Jakob disease, traumatic brain dementia, other physical and chemical factors (such as drugs, alcohol, CO), systemic disease (hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial occupation (a subdural hematoma, brain tumor), the endocrine system disease (thyroid disease, parathyroid disease), and vitamins deficiency or any other causes of dementia
2. The history of nervous system diseases, including stroke, optic myelitis, Parkinson's disease, epilepsy, etc
3. Psychiatric patients, including schizophrenia or other mental illnesses, bipolar disorder, major depression, or delirium
4. There are unstable or serious heart, lung, liver, kidney, endocrine, and hematopoietic system diseases, or Poor prognosis because of malignant diseases such as tumors.
5. Vision or hearing problems that lead to poor performance on cognitive tests
6. Two years history of severe alcoholism, and drug abuse
7. Participants who participated in any other trial 30 days prior to their screening visit
8. Contraindication of MRI scanning
9. Special requirements for diet, e.g., allergy to common food or on a special diet due to medical needs
10. Participants who cannot be followed for at least 6 months (due to a health situation or migration)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline global cognitive function at one year | One year
  Change from baseline general cognitive performance at one year assessed by Mini-mental state examination (MMSE)
Change from baseline memory at one year | One year
  Change from baseline verbal memory using the Auditory verbal learning test (AVLT)
Change from baseline visual spatial ability and visual memory at one year | One year
  Change from baseline visual spatial ability and visual memoryevaluated by the Rey-Osterrieth complex figure test (CFT)

SECONDARY OUTCOMES:
Changes in cognition assessed by Clock drawing test, Symbol-digit test, Trail making test, Boston naming test and Language fluency test | One year
  Executive function
Changes in hippocampus related neural circuit-specific resting-state connectivity (FC) | One year
  Neural connectivity by functional MRI
Changes in structural brain MRI including volume of hippocampus and other specific brain regions | One year
  Brain structure by MRI
Changes in Inflammatory biomarkers | One year
  Serum interleukins and tumor necrosis factors
Changes in gut microbiota | One year
  Number of genera and abundance of microbiota in feces and blood
Changes in Metabolic biomarkers | One year
  Low-density lipoprotein, high-density lipoprotein, and total cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No